CLINICAL TRIAL: NCT00043914
Title: A Multicenter, Open-Label Conversion of Valproate Monotherapy to Lamotrigine Monotherapy in Patients With Epilepsy
Brief Title: Measurement Of Serum Levels Of Two Antiepileptic Drugs During Conversion In Patients With Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAM40013
Record Dates: First submitted 2002-08-14; First posted 2002-08-16 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Epilepsy
Keywords: epilepsy; monotherapy conversion
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

INTERVENTIONS:
Drug: lamotrigine

SUMMARY:
This study includes patients 16 years of age or older with a confident diagnosis of epilepsy who are currently treated with an antiepileptic drug (AED) monotherapy but require a change in therapy due to inadequate seizure control and/or unacceptable side effects.

ELIGIBILITY:
INCLUSION CRITERIA:

* 16 years old or older.
* Have confident diagnosis of epilepsy.
* Have been on the medication valproate for at least 3 months and is currently on a stable daily dose.
* Male or female; females of child-bearing potential must have negative pregnancy test at screen and must agree to use an acceptable birth control method.

EXCLUSION CRITERIA:

* A history of hypersensitivity to the drug being studied.
* Currently being treated with or has been treated in the past with the drug being studied.
* Undergoing polytherapy treatment with the medication valproate and one or more other antiepileptic drug(s).
* If undergoing treatment with vagal nerve stimulation, has had device implanted more than 30 days prior to enrollment.
* Has taken an investigational drug or the medication Felbatol within the previous 30 days.
* Is abusing alcohol and/or other substances.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72
Dates: Start 2002-01-14 (Actual); Primary Completion 2003-01-29 (Actual); Study Completion 2003-01-29 (Actual)

PRIMARY OUTCOMES:
Drug levels of lamotrigine.

SECONDARY OUTCOMES:
This study has no secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Sale ME, Natarajan S, Biton V, Vuong A, Hammer AE, Messenheimer JA, Blum D. A dosing algorithm for converting from valproate monotherapy to lamotrigine monotherapy in patients with epilepsy. Epilepsy Behav. 2005 Feb;6(1):63-70. doi: 10.1016/j.yebeh.2004.11.002. PMID 15652736
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: LAM40013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LAM40013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LAM40013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LAM40013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LAM40013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LAM40013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LAM40013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register